CLINICAL TRIAL: NCT06896773
Title: Effect of Training in Normobaric Hypoxia on Cardiac Markers
Acronym: HYPO-CARDIAC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NdS-II/SP/0431/2024/01; NdS-II/SP/0431/2024/01 (Other Grant/Funding Number: Ministry of Science and Higher Education of Poland)
Record Dates: First submitted 2025-01-09; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Heart Disease
Keywords: normobaric hypoxia; cardiac markers; endurance training; resistance training
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Trained group - cyclists and triathletes (Experimental): The participants in training group will meet the following criteria: male, aged 20-40, VO2max of not less than 60 ml/kg/min, training experience of at least 6 years and at least a six-month wash-out period from any previous altitude training. Additionally, inclusion criteria in both groups will be: no chronic diseases; (3) systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. The study will exclude participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
  Interventions: Other: Impact of Normobaric Hypoxia on Cardiac Biomarkers in trained men
- Untrained group - healthy men (Experimental): Inclusion criteria will be: male, aged 20-40 years, no chronic diseases, systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. The study will exclude participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
- LHTL group (live high, train low) (Experimental): The LHTL group: male, aged 20-40, competitive cyclists in the pre-competition phase of training, with a wash-out period of at least six months after previous altitude training, VO2max of not less than 60 ml/kg/min, training experience of at least 6 years, no chronic diseases, systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. The LHTL group will be exposed to normobaric hypoxia (FIO2 = 14.4%, corresponding to an altitude of 3000 m a.s.l.) in a hotel room for 11 to 12 hours a day (evenings and nights) and train under normoxic conditions.The study will exclude participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
- IHT group- intermittent hypoxic training (Experimental): Participants in the IHT group: male, aged 20-40, competitive cyclists in the pre-competition phase of training, with a wash-out period of at least six months after previous altitude training, VO2max of not less than 60 ml/kg/min, training experience of at least 6 years, no chronic diseases, systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. Participants in the IHT group will live in normoxic conditions, but part of their training will be performed in normobaric hypoxia (FIO2 = 14.4%, 3000 m a.s.l.) in a hypoxic chamber. The study will exclude participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
  Interventions: Other: Effects of Hypoxic Endurance Training on Cardiac Biomarkers in the IHT group
- Control group - C (Experimental): The C group: male, aged 20-40, competitive cyclists, in the pre-competition phase of training, with a wash-out period of at least six months after previous altitude training, VO2max of not less than 60 ml/kg/min, training experience of at least 6 years, no chronic diseases; systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. The participants will live and perform endurance training in normoxic conditions. The study will exclude participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
  Interventions: Other: Effects of Hypoxic Endurance Training on Cardiac Biomarkers in the Control group
- HRT group - hypoxic resistance training (Experimental): The participants in the HRT group: male, aged 20-40, at least three years of systematic strength training, wash-out period of at least six months after previous altitude/hypoxic training, no chronic diseases, systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. Participants will perform resistance training in normobaric hypoxia (FIO2 = 14.4%, 3000 m a.s.l.). The study will be excluded participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
  Interventions: Other: Effects of Hypoxic Strength Training on Cardiac Biomarkers in the HRT group
- NRT group - normoxia resistance training (Experimental): The participants in the NRT group: male, aged 20-40, at least three years of systematic strength training, wash-out period of at least six months after previous altitude/hypoxic training, no chronic diseases, systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg. Participants will perform resistance training in normoxia. The study will be excluded participants who use drugs, drink alcohol or smoke, have hypertension, prematurely stopped the exercise test.
  Interventions: Other: Effects of Hypoxic Strength Training on Cardiac Biomarkers in the NRT group

INTERVENTIONS:
Other: Impact of Normobaric Hypoxia on Cardiac Biomarkers in trained men — The intervention will consist of three series differing in terms of simulated altitude: S1 (normoxia), S2 (2000 m a.s.l.), and S3 (3000 m a.s.l.). Each research series will consist of one day of the measurements. All participants will perform two ergocycle tests (the graded exercise test GXT and constant-workload exercise test CXT at the individual lactate threshold workload (WRLT) until volitional exhaustion) with 10 minutes of active recovery break in different environment (S1, S2, S3- 3000). The order of the series will be randomized across all participants. The fraction of inspired oxygen (FIO2) will depend on the series and will be as follows: S1 (normoxia) = 20.9%; S2 (2000 m a.s.l.) = 16,5%; S3 (3000 m a.s.l.) = 14.4%. The hypoxic environment will be maintained using AirZone climate technology (AirSport). Between the series, there will be a one-week active rest break excluding exposure to hypoxia and performance of high-intensity exercise.
  Arms: Trained group - cyclists and triathletes
Other: Effects of Hypoxic Endurance Training on Cardiac Biomarkers in the IHT group — The participants in IHT group will live in normoxic conditions, but part of their training will be performed in normobaric hypoxia in a hypoxic chamber. The experiment will consist of two series of testing: S1 (baseline) and S2 (after 3 weeks of training and 3 days of rest). All participants will perform the same testing protocol as in stage 1-albeit in a normoxic environment and after 72h of rest, all testing procedures will be repeated in a hypoxic environment.
  Arms: IHT group- intermittent hypoxic training
Other: Effects of Hypoxic Strength Training on Cardiac Biomarkers in the NRT group — The participants in the NRT group will perform resistance training in normoxia. The experiment will consist of two series of testing (S1 and S2), performed in a laboratory. S1 will involve baseline testing, while S2 will be performed after three weeks of training after 3 days of rest. Each research series will consist of three measurement days. The testing protocol and blood sampling will be the same as in the first and second stages of the research. After next 72h of rest, all participants will have their muscle strength assessed using the one-repetition maximum (1RM) test in normoxia environment. The tests will be conducted in two exercises: a barbell bench press and a barbell squat.
  Arms: NRT group - normoxia resistance training
Other: Impact of Normobaric Hypoxia on Cardiac Biomarkers in untrained men — The intervention will consist of three series differing in terms of simulated altitude: S1 (normoxia), S2 (2000 m a.s.l.), and S3 (3000 m a.s.l.). Each research series will consist of one day of the measurements. All participants will perform two ergocycle tests (the graded exercise test GXT and constant-workload exercise test CXT at the individual lactate threshold workload (WRLT) until volitional exhaustion) with 10 minutes of active recovery break in different environment (S1, S2, S3- 3000). The order of the series will be randomized across all participants. The fraction of inspired oxygen (FIO2) will depend on the series and will be as follows: S1 (normoxia) = 20.9%; S2 (2000 m a.s.l.) = 16,5%; S3 (3000 m a.s.l.) = 14.4%. The hypoxic environment will be maintained using AirZone climate technology (AirSport). Between the series, there will be a one-week active rest break excluding exposure to hypoxia and performance of high-intensity exercise.
Other: Effects of Hypoxic Endurance Training on Cardiac Biomarkers in the LHTL group — The participants from the LHTL group will be exposed to normobaric hypoxia (FIO2 = 14.4%, corresponding to an altitude of 3000 m a.s.l.) in a hotel room for 11 to 12 hours a day (evenings and nights). Participants in this group will perform interval training under normoxic conditions. The experiment will consist of two series of testing: S1 (baseline) and S2 (after 3 weeks of training and 3 days of rest). All participants will perform the same testing protocol as in stage 1-albeit in a normoxic environment and after 72h of rest, all testing procedures will be repeated in a hypoxic environment.
Other: Effects of Hypoxic Endurance Training on Cardiac Biomarkers in the Control group — The participants in the C group will live and train in normoxic conditions. The experiment will consist of two series of testing: S1 (baseline) and S2 (after 3 weeks of training and 3 days of rest). All participants will perform the same testing protocol as in stage 1-albeit in a normoxic environment and after 72h of rest, all testing procedures will be repeated in a hypoxic environment.
  Arms: Control group - C
Other: Effects of Hypoxic Strength Training on Cardiac Biomarkers in the HRT group — The participants in the HRT group will perform resistance training in normobaric hypoxia (FIO2 = 14.4%, 3000 m a.s.l.). The experiment will consist of two series of testing (S1 and S2), performed in a laboratory. S1 will involve baseline testing, while S2 will be performed after three weeks of training after 3 days of rest. Each research series will consist of three measurement days. The testing protocol and blood sampling will be the same as in the first and second stages of the research. After next 72h of rest, all participants will have their muscle strength assessed using the one-repetition maximum (1RM) test in normoxia environment. The tests will be conducted in two exercises: a barbell bench press and a barbell squat.
  Arms: HRT group - hypoxic resistance training

SUMMARY:
The goal of this study is to determine changes in the concentration of cardiac biomarkers in blood in response to a single bout of exercise performed until volitional exhaustion under hypoxic conditions, and in response to endurance and resistance training in athletes in hypoxia. The investigators hypothesize that: (1) adverse changes in the myocardium may occur during exercise in acute normobaric hypoxia, but they are at least partially reversed by adaptive alterations induced by training in hypoxia; (2) this response is identical in athletes with eccentric cardiac hypertrophy and those with concentric cardiac hypertrophy.

The study consists of three stages. Stage 1 (completed) has examine changes in the blood levels of cardiac biomarkers in response to a single bout of exercise performed until volitional exhaustion in normoxia and during different levels of hypoxia (2000, 3000m). This stage has examined men aged 20-40 years involved in competitive cycling and triathlon, and untrained, healthy men.

Stage 2 of the study will examine changes in the blood levels of cardiac biomarkers in cyclists (aged 20-40) in response to a 3-week endurance training in hypoxia and to passive prolonged exposure (11 to 12 hours a day) to a simulated altitude of 3000m. Stage 3 will examine changes in blood levels of cardiac biomarkers in response to a 3-week resistance training in hypoxia (3000m). This stage of the study will involve men aged 20-40 training in strength sports.

The project will help clarify the effects of hypoxia on the physiological state of the heart in athletes with eccentric or concentric cardiac hypertrophy, as well as determine the differences between competitive athletes vs. untrained, healthy men in the response to hypoxia. The findings may be used in planning and controlling the training process in both strength and endurance disciplines. The research to be conducted in the project is basic research, but it may have a certain applicative aspect.

DETAILED DESCRIPTION:
The goal of this interventional trial is to determine changes in the concentration of cardiac biomarkers in blood in response to exercise performed until volitional exhaustion: (1) after a single exposure to normoxia and normobaric hypoxic conditions with varying levels of the hypoxic stimulus, in trained and untrained men; (2) after 3 weeks of endurance training in normobaric hypoxia in cyclists (eccentric hypertrophy); (3) after 3 weeks of resistance training in normobaric hypoxia in strength athletes (concentric hypertrophy).

The research project involves assessing the physiological state of the myocardium after acute and chronic exposure to normobaric hypoxia in athletes with eccentric and concentric cardiac hypertrophy by measuring selected cardiac biomarkers in blood serum: cardiac troponins I and T (cTnI and cTnT), myoglobin (Myo), and the creatine kinase-myocardial band fraction (CK-MB), B-type natriuretic peptide (NT-proBNP), N-terminal pro-hormone of BNP (H-FABP) and ischemia-modified albumin (IMA). In addition, the levels of the following markers will be observed: hypoxia-inducible factor-1 (HIF-1α), vascular endothelial growth factor A (VEGF-A), nitrites and nitrates (NO breakdown products).

The study consists of three stages. Stage 1 (has been completed). All participants have performed two consecutive ergocycle tests (the graded exercise test GXT and constant-workload exercise test CXT with 10 minutes of active recovery break in different environment (S1-normoxia, S2-2000 m a.s.l., S3- 3000 m a.s.l.). The fraction of inspired oxygen (FIO2) is as follows: S1 (normoxia) = 20.9%; S2 (2000 m a.s.l.) = 16,5%; S3 (3000 m a.s.l.) = 14.4%. The hypoxic environment was maintained using AirZone climate technology (AirSport).

In stage 2 of the study, changes in the blood levels of cardiac biomarkers in 36 male cyclists in response to 3 weeks of endurance training in hypoxia (3000m) will be examined. The participants will be randomly assigned to three groups: (1) LHTL "live high, train low"; (2) IHT "intermittent hypoxic training"; (3) the control group (C) - normoxic training.

The experiment will consist of two series of testing: S1 (baseline tests) and S2 (tests after three weeks of training and after 3 days of rest).

All athletes will be trained at a professional training center providing enough hypoxic hotel rooms and training chambers. The participants will be provided with standardized meals and snacks. The training load will be recorded using the power meters (Vector, Garmin), and the obtained data will be analyzed with the software WKO5 (TrainingPeaks). All athletes will follow the same training regimen for three weeks (three basic microcycles and three days of recovery). Exercise intensity will be individually adjusted according to the lactate threshold workload (WRLT) of each athlete. In each training microcycle, all participants will perform three interval training sessions in laboratory conditions (a hypoxic chamber). Each interval training session will start with a 15-minute warm-up, followed by 50-60 minutes of the main exercise, and a 10-minute cooldown. The warm-up will be performed at the intensity of 60-80% WRLT/WRLThyp. In the main part, the participants will perform 4-5 intervals lasting 4-5 minutes with a workload of 110% WRLT/WRLThyp. The recovery period between intervals will last 6-8 min with a workload of 70% WRLT/WRLThyp. The cooldown phase will consist of 10 minutes of continuous exercise with a workload of 60% of WRLT/WRLThyp.

Stage 3 changes in blood levels of cardiac biomarkers in 28 men strength athletes in response to 3 weeks of resistance training in hypoxia (3000m) will be examined. The participants will be randomized into two equal groups: hypoxic resistance training (HRT) and normoxic resistance training (NRT). The participants in the HRT group will perform resistance training in normobaric hypoxia (FIO2 = 14.4%, 3000 m a.s.l.), while the participants in the NRT group will perform the same training, but in normoxia. The experiment in stage 3 will consist of two series of testing (S1 and S2), performed in a laboratory. Each research series will consist of three measurement days. On the first day, all participants will perform two consecutive ergocycle tests with 10 minutes of active recovery break in normoxia environment. The testing protocol and blood sampling will be the same as in the first and second stages of the research. After 72h of rest, participants will repeat the entire testing protocol under hypoxic conditions. The order of the conditions (hypoxia vs. normoxia) will be randomized across all participants. After next 72h of rest, all participants will have their muscle strength assessed using the one-repetition maximum (1RM) test in normoxia environment. The tests will be conducted in two exercises: a barbell bench press and a barbell squat. Maximum muscle strength will be measured using the following protocol: 10 min warm-up, the 1RM test- a maximum of four consecutive attempts with increasing workloads and a five-minute rest period between attempts, selection of the first workload - 70% of the participant's assumed strength capacity. Weight will gradually increased by approximately 2.5-20 kg until the participant is unable to complete the repetition. The participant's final 1RM is the last-attempt workload performed at full range and with constant speed.

Both groups (HRT and NRT) will follow the same training protocol. All training sessions will be performed in a normobaric hypoxic chamber and participants will not be informed about the conditions in the chamber. The resistance training will consist of three training sessions per week. Each unit will consist of a 15-minute warm-up and a 50-minute main part. In the main part, the participants will perform barbell bench presses and barbell squats. For each exercise, they will perform eight sets of 10 repetitions with a workload of 70% 1RM. The passive recovery period between the sets will be three minutes. In all groups, the workload will be increased individually by 5 kg if the participant performs all scheduled repetitions twice in a row (160).

For each participant in all series of testing (stage 1, 2, and 3), blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT) tests, after 2, 6, and 24 hours. The order of conditions (normoxia vs. hypoxia) in all series of testing will be randomized across all participants, and all series of testing and training sessions will be performed in a normobaric hypoxic chamber (AirZone, AirSport). Participants will not be informed about the conditions. Throughout the research project, all participants will be on a controlled mixed diet and will not be supplemented.

Testing protocol in all stages of the research project In all series of testing, before breakfast, body mass and body composition will be taken between 7 and 7:30 am. Body height will be measured using an anthropometer with an accuracy of 0.5 cm, and body composition will be estimated using bioelectrical impedance analysis (InBody 220, Biospace).

Then, two hours after the consumption of a light mixed meal (5 kcal/1kg body weight; 50% carbohydrates, 30% fat, 20% protein), all participants will perform two consecutive ergocycle tests with 10 minutes of active recovery break. The all tests will be performed on a cycle ergometer (Excalibur Sport, Lode BV) adjusted individually to each participant.

The first test will be included the graded exercise test (GXT) until volitional exhaustion. The exercise will start with a workload of 90 W, with increments of 30 W every three minutes until volitional exhaustion. At rest (3 minutes before the test) and during the GXT, continuous recording of heart rate (HR) and minute ventilation (VE), breathing frequency (BF), oxygen uptake (VO2) and expired carbon dioxide (VCO2), and end-tidal oxygen tension (PETO2) and end-tidal carbon dioxide tension (PETCO2) will be performed by means of a fast gas analyser (MetaLyzer 3B, Cortex) using the breath-by-breath method. The following criteria will be used to assess the VO2max: (1) stabilization of VO2 despite a further increase in load (ΔVO2<150mL/min), (2) gradual decrease in peak VO2 during maximal load. Additionally, at rest and during the GXT, continuous recording of blood oxygen saturation (SpO2) will be measured (WristOx2, Nonin Medical Inc.).

In the case of the last uncompleted stage, maximal workload (WRmax) will be calculated from the following formula: WRmax=WRk+ (t/T x WRp), where WRk = previous workload, t = exercise duration with the work-load until premature failure, T = duration of each workload, WRp = the amount of workload by which exercise intensity increased during the test. Cardiac output (Q) will estimate by VO2max, and will calculated by the following formula: Q= 100 x VO2/(5.72 + 10.5 x VO2/VO2max) using MetaSoft Studio (Cortex, Germany). Stroke volume (SV) will calculate as follows: SV= Q/HR At the end of each load (last 15 s) capillary blood samples will be obtained from fingertips in order to determine blood lactate levels (LA; SUPER GL2, Dr. Müller Gerätebau GmbH). These data will be used to analyse the kinetics of LA concentration in blood, evaluate individual anaerobic threshold based on the Dmax method. Furthermore, before and immediately after completion of the GXT, capillary blood will be obtained from the fingertip to determine the acid-base balance and to analyse selected gas exchange indicators: oxygen saturation (SaO2), partial pressure of oxygen (pO2) and partial pressure of carbon dioxide (pCO2) in the blood (OPTI CCA-TS2 Blood Gas and Electrolyte Analyzer, OPTI Medical Systems). This will be followed by a 10-minute active rest break (30% of the maximum workload reached during the test until volitional exhaustion, WRmax).

Then, the participants will perform constant-workload exercise test (CXT) at the individual lactate threshold workload (WRLT) until volitional exhaustion. During the CXT, the participants will be allowed to drink water ad libitum. Before and immediately after completion of the CXT, capillary blood will be obtained from the fingertip to determine the LA concentration and acid-base balance. Additionally, at rest and during the CXT, continuous recording of HR and SpO2 will be measured (WristOx2, Nonin Medical Inc.). In all series of tasting during each stage of the research project, participants will undergo 2 complete Transthoracic Echocardiography (TTE) examinations using a GE Medical System Vivid 7 with a 2.5-MHz transducer by the same investigator. M-mode, two-dimensional imaging, and Doppler techniques will be performed.

For each participant, blood samples of 8mL will be taken from the antecubital vein at six time points during each series of the study: before and immediately after GXT+CXT tests, after 2, 6, and 24 hours. Blood morphology will be assessed in EDTA-anticoagulated venous blood on an automated hematology analyzer (model ADVIA 60). The levels of cTnI and cTnT, NT-proBNP, H-FABP, IMA, HIF-1α, VEGF-A will be determined using commercially available ELISA kits according to the manufacturer's instruction. Serum activities of CK-MB will be measured calorimetrically with the use of commercial kits. Serum NO2- and/or NO3- levels will be determined calorimetrically with the use of commercial kits employing the Griess method, with and without enzymatic conversion of NO3- into NO2-.

ELIGIBILITY:
Inclusion Criteria:

* males
* age 20-40 years
* VO2max of not less than 60 ml/kg/min
* training experience of at least 6 years (for stage 1) and 3 years (for stage 2 and 3)
* at least a six-month wash-out period from any previous altitude training, - competitive cyclists in the pre-competition phase of training (for stage 2)
* no chronic diseases
* systolic blood pressure 100-140 mmHg and diastolic blood pressure 60-90 mmHg.

Exclusion Criteria:

* participants who use drugs
* drink alcohol or smoke,
* hypertension
* prematurely stopped the exercise test.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine blood profile based on complete blood count (CBC) [million/mm3]
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine HIF-1α [%oxygen].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine VEGF-A [pg/ml].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine cTnI [ng/L] and cTnT [ng/L].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine Myo [mcg/L].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine CK-MB [IU/L].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine H-FABP [ng/mL].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine IMA [U/L].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine NT-proBNP [pg/mL].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine nitrites and nitrates [mg/l].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on myocardial contractility in trained and untrained men. | Up to 1 year
  For each participant, before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours echocardiography will undergo.
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine VO2max [ml oxygen/kg of body weight/minute].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine complete blood count (CBC) [million/mm3].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine HIF-1α [%oxygen].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine VEGF-A [pg/ml]..
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine cTnI [ng/L] 5 and cTnT [ng/L].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine Myo [mcg/L].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine H-FABP [ng/mL].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine IMA [U/L].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine NT-proBNP [pg/mL].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine nitrites and nitrates [mg/l].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine VO2max [ml oxygen/kg of body weight/minute].
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine acid-base balance [-].
To determine the relationship between the fitness level (trained vs. untrained) and changes in myocardial contractility in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Echocardiography at rest and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, will undergo.
To evaluate the muscle strength in normoxia | Up to 2 years
  Muscle strength [1RM] test in normoxia environment. The tests will be conducted in two exercises: a barbell bench press and a barbell squat.
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on myocardial contractility in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, echocardiography at rest and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will undergo.
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine complete blood count (CBC) [million/mm3].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine HIF-1α [%oxygen].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine VEGF-A [pg/ml].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine cTnI [ng/L] and cTnT [ng/L].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine Myo [mcg/L].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine CK-MB [IU/L].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine H-FABP [ng/mL].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine IMA [U/L].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine NT-proBNP [pg/mL].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine nitrites and nitrates [mg/l].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine VO2max [ml oxygen/kg of body weight/minute].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine LA concentration [mmol/L].
To evaluate the effect of 3 weeks of endurance training in two methods of hypoxic training (LH-TL, and IHT) on cardiac biomarkers in response to a single exercise until volitional exhaustion in normoxia and hypoxia | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine acid-base balance [-].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT) tests, after 2, 6, and 24 hours. The blood samples will be used to determine complete blood count (CBC) [million/mm3].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine HIF-1α [%oxygen].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine VEGF-A [pg/ml].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine cTnI [ng/L] and cTnT [ng/L].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine Myo [mcg/L].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine CK-MB [IU/L].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine H-FABP [ng/mL].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine IMA [U/L].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine NT-proBNP [pg/mL].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine nitrites and nitrates [mg/l].
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine VO2max [ml oxygen/kg of body weight/minute]
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine LA concentration [mmol/L]
To evaluate the effect of 3 weeks of resistance training in hypoxia on cardiac biomarkers concentration in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine acid-base balance [-].
To evaluate the effect of 3 weeks of resistance training in hypoxia on myocardial contractility in response to a single exercise until volitional exhaustion in normoxia and hypoxia (3000 m. a.s.l) | Up to 2 years
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT) tests, after 2, 6, and 24 hours. Echocardiography at rest and immediately the tests will undergo.
To determine the relationship between the fitness level (trained vs. untrained) and changes in cardiac biomarker concentrations in blood in response to a single exercise until volitional exhaustion in normoxia and hypoxia. | Up to 1 year
  Changes in the concentration of cardiac biomarkers in blood in response to two consecutive ergocycle tests during exposure normoxia and different levels of hypoxia in trained and untrained man during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours will be measured. The blood samples will be used to determine CK-MB [IU/L].
The effect of single exercise until volitional exhaustion in normoxia and normobaric hypoxic conditions, on cardiac biomarker concentrations in blood in trained and untrained men. | Up to 1 year
  For each participant, blood samples will be taken at five time points during each series of the study: before and immediately after the graded exercise test (GXT) and constant-workload exercise test (CXT), after 2, 6, and 24 hours. The blood samples will be used to determine acid-base balance [-].

CONTACTS AND LOCATIONS:
Overall Officials: Miłosz Czuba, Prof., Study Chair — Józef Piłsudski University of Physical Education in Warsaw, Poland
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Poland, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Additional supporting information will be available upon request.

REFERENCES:
- [Derived] Robert G, Milosz C, Kamila P, Ewa K, Adam N, Michal S, Natalia GZ, Katarzyna K, Jozef L. The Impact of High-Intensity Exercise in Normobaric Hypoxia on Right Ventricular Function in Trained and Untrained Men-An Echocardiographic Study. Compr Physiol. 2026 Feb;16(1):e70090. doi: 10.1002/cph4.70090. PMID 41496576